CLINICAL TRIAL: NCT01579071
Title: A Randomized, Controlled, Double-blind Trial of the Efficacy and Safety of CO2 vs Room Air Insufflation During ESD for Gastric Tumor
Brief Title: Efficacy and Safety of CO2 vs Room Air Insufflation During ESD for Gastric Tumor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Ju Seung Kim, MD, principle investigator, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GIRBA2681-2012
Record Dates: First submitted 2012-04-05; First posted 2012-04-17 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Gastric Tumor
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CO2 sufflation group (Experimental)
  Interventions: Procedure: CO2 or room air insufflation during ESD for gastric tumor
- Room air sufflation group (Experimental)
  Interventions: Procedure: CO2 or room air insufflation during ESD for gastric tumor

INTERVENTIONS:
Procedure: CO2 or room air insufflation during ESD for gastric tumor — CO2 insufflation group : CO2 will be insufflated via the endoscope during procedure as needed, Room air insufflation group : Room air will be insufflated via the endoscope during procedure as needed

SUMMARY:
Insufflation is essential procedure to observe the lumen of gastrointestinal tract in gastroscopy or colonoscopy Currently, most of hospital in Korea are using room air for insufflation According to recent clinical studies have shown that carbon dioxide have better safe and reduce stomachache than room air when endoscopy and endoscopic procedure is performed.

However, there was still no research data or study in Korea. In this study, the investigators will try to make comparison between Carbon dioxide and room air insufflation for endoscopic submucosal dissection for Gastric Tumor and investigate the efficacy and safety

ELIGIBILITY:
Inclusion Criteria:

* Patients who have gastroscopy and colonoscopy or ESD for gastric tumor under sedation in department of gastroenterology, Gachon University Gil Medical Center

Exclusion Criteria:

* Age : < 19 years old
* Underlying disease : COPD requiring O2
* Known CO2 retention
* Opiate abuse for chronic pain
* Nonreader or short in understanding
* Pregnancy
* Any medical instabilities expected to not be in safe

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Abdominal pain related to each insufflation | 1 day
  Patients will be received questionnaire (100mm visual analogue scale, VAS) and record their score in 0, 1, 3, 6, 24 hours after endoscopic procedure.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 1 day
  The investigators will check the side effect during and after pocedure. If any side effect occur, the investigators will stop the procedure and act right away.

CONTACTS AND LOCATIONS:
Locations (1):
- Gachon University Gil Medical Center Department of Gastroentorology, Incheon, Incheon, South Korea

REFERENCES:
- [Derived] Kim SY, Chung JW, Park DK, Kwon KA, Kim KO, Kim YJ. Efficacy of carbon dioxide insufflation during gastric endoscopic submucosal dissection: a randomized, double-blind, controlled, prospective study. Gastrointest Endosc. 2015 Dec;82(6):1018-24. doi: 10.1016/j.gie.2015.05.043. Epub 2015 Jul 2. PMID 26142555